CLINICAL TRIAL: NCT04628273
Title: A Prospective Cohort Study of Large Pancreatic Radiolucent Stone
Brief Title: Treatment Strategy of Pancreatic Radiolucent Stone
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology，Changhai Hospital；Academician of Chinese Academy of Engineering, Changhai Hospital
Other Study IDs: Large PRS
Record Dates: First submitted 2020-11-07; First posted 2020-11-13 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Lithotripsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- radiolucent stone group
  Interventions: Procedure: encoscopic retrograde cholangio-pancreatography, extracorporeal shock wave lithotripsy
- radiopaque stone group
  Interventions: Procedure: encoscopic retrograde cholangio-pancreatography, extracorporeal shock wave lithotripsy

INTERVENTIONS:
Procedure: encoscopic retrograde cholangio-pancreatography, extracorporeal shock wave lithotripsy

SUMMARY:
Treatment strategy of chronic pancreatitis (CP) patients with large pancreatic radiolucent stone (≥ 5mm) has not been established. We aimed to figure out clinical features and efficacy of endotherapy for large pancreatic radiolucent stone.

DETAILED DESCRIPTION:
1. Treatment strategy of CP patients with large pancreatic stone：

1. . For patients with large radiolucent stone，ERCP with balloon sphincteroplasty was performed directly to remove radiolucent stone. If ERCP intubation failed, endoscopic ultrasound-guided drainage of pancreatic duct, surgery or medication would be applied. ESWL was performed in the following situations. Frist, MPD strictures was so severe that dilation catheter can not be inserted during ERCP. Second, there was cystic dilatation in MPD and pancreatic radiolucent stone located in cystic dilatation could not be extracted by extraction balloon or basket. In the above cases, the naso-pancreatic catheterwas inserted during ERCP, and then ESWL would be performed with repeated injection of contrast medium. After ESWL, repeated washing and negative pressure drainage were performed, and at last contrast medium was injected again to make sure the stones were cleared. For patients without MPD strictures, the nasopancreatic catheter can be directly removed, otherwise the nasopancreatic duct would be cut off into a stent.
2. . For patients with large radiopaque stone, repeated P-ESWL sessions were performed, and ERCP was routinely performed 48 hours after the last P-ESWL. If ERCP intubation failed, medication or surgery would be recommended.

2. A prospective cohort study was conducted in CP patients with large radiolucent stone. Patients with large radiopaque stone were matched as the control group, with a ratio of 1:2 according to admission time.

3. The primary outcome was pain relief. The secondary outcomes were stone clearance, quality of life score, and changes in pancreatic exocrine and endocrine function.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of chronic pancreatitis; With pancreatic radiolucent stones large than 5mm

Exclusion Criteria:

Autoimmune pancreatitis; Groove pancreatitis; Pancreatic cancer diagnosed within 2 years after diagnosis of chronic pancreatitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CP patients with pancreatic radiolucent stones large than 5mm from March 2011 to December 2018 admitted to Changhai Hospital were included in this study. Patients with pancreatic radiopaque stones large than 5mm were matched as the control group, with a ratio of 1:2 according to admission time. CP was diagnosed primarily based on the Asia-Pacific consensus. Pancreatic radiopaque stone was diagnosed by CT scan while radiolucent stone by MRI or MRCP.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
rate of pain relief | after treatment to 2020-01-30
  Pain relief is evaluated by Izbicki pain score and classified as complete relief (Izbicki pain score ≤ 10) or partial relief (Izbicki pain score > 10 after a decrease of > 50%)

SECONDARY OUTCOMES:
rate of stone clearance | during ERCP procedure
  Rate of stone clearance is evaluated by ERCP as follows: a) complete clearance as clearance of > 90% of stone volume; b) partial clearance as clearance of 50%-90% of stone volume; c) unsuccessful clearance as less than 50% clearance of stone volume
score of life quality | after treatment to 2020-01-30
  Quality of life score was a subjective evaluation index of patient which ranged from 0 to 100, with higher score indicating a better quality of life

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tandan M, Reddy DN, Santosh D, Vinod K, Ramchandani M, Rajesh G, Rama K, Lakhtakia S, Banerjee R, Pratap N, Venkat Rao G. Extracorporeal shock wave lithotripsy and endotherapy for pancreatic calculi-a large single center experience. Indian J Gastroenterol. 2010 Jul;29(4):143-8. doi: 10.1007/s12664-010-0035-y. Epub 2010 Aug 18. PMID 20717860
- [Background] Neuhaus H. Fragmentation of pancreatic stones by extracorporeal shock wave lithotripsy. Endoscopy. 1991 May;23(3):161-5. doi: 10.1055/s-2007-1010647. No abstract available. PMID 1860446
- [Background] Sauerbruch T, Holl J, Sackmann M, Paumgartner G. Extracorporeal lithotripsy of pancreatic stones in patients with chronic pancreatitis and pain: a prospective follow up study. Gut. 1992 Jul;33(7):969-72. doi: 10.1136/gut.33.7.969. PMID 1644340
- [Background] Delhaye M, Arvanitakis M, Verset G, Cremer M, Deviere J. Long-term clinical outcome after endoscopic pancreatic ductal drainage for patients with painful chronic pancreatitis. Clin Gastroenterol Hepatol. 2004 Dec;2(12):1096-106. doi: 10.1016/s1542-3565(04)00544-0. PMID 15625655
- [Background] Maydeo A, Bhandari S, Bapat M. Endoscopic balloon sphincteroplasty for extraction of large radiolucent pancreatic duct stones (with videos). Gastrointest Endosc. 2009 Oct;70(4):798-802. doi: 10.1016/j.gie.2009.05.004. PMID 19788986